CLINICAL TRIAL: NCT02524756
Title: Feasibility and Functional Outcome of Laparoscopic Nerve Sparing Radical Hysterectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Osama Mohammad Ali ElDamshety (Other)
Collaborators: Catholic University of the Sacred Heart (Other)
Responsible Party: Sponsor-Investigator, Osama Mohammad Ali ElDamshety, surgical oncology, Mansoura University
Organization: Mansoura University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LNS-RH
Record Dates: First submitted 2015-08-12; First posted 2015-08-17 (Estimated); Last update posted 2018-03-06 (Actual); Status verified 2018-03

CONDITIONS: Cervical Cancer
Keywords: nerve sparing radical hysterectomy
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group (A) (Active Comparator): laparoscopic nerve sparing radical hysterectomy type III/C1
  Interventions: Procedure: laparoscopic nerve-sparing radical hysterectomy-type III/C1
- Group (B) (Active Comparator): laparoscopic radical hysterectomy type III/C2
  Interventions: Procedure: laparoscopic radical hysterectomy (type III/C2).

INTERVENTIONS:
Procedure: laparoscopic nerve-sparing radical hysterectomy-type III/C1
  Arms: Group (A)
Procedure: laparoscopic radical hysterectomy (type III/C2).
  Arms: Group (B)

SUMMARY:
The aim of this study is to assess:

1. Evaluation of the feasibility of laparoscopic nerve sparing radical hysterectomy type III/C1 as regard surgical technique, blood loss and operative time.
2. Evaluate patients' outcome as regard bladder function.

in order to preserve the function of the bladder and the rectum, it is necessary to modify the traditional procedures, so as to identify the precise anatomical information directing the technique for optimal preservation of bladder function at the time of radical hysterectomy.

The laparoscopic technique offers several well-known advantages. Under the magnified view of the laparoscope, the anatomy can be clearly visualized to allow for the meticulous and precise dissection of the para-cervical structures and areolar tissue, including the blood vessels and the nerves.

Laparoscopic identification (neurolysis) of the inferior hypogastric nerve and inferior hypogastric plexus is a feasible procedure for trained laparoscopic surgeons who have a good knowledge not only of the retroperitoneal anatomy but also of the pelvic neuro-anatomy as this qualification could prohibit long-term bladder and voiding dysfunction during nerve-sparing radical hysterectomy

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years.
2. Karnofsky > 80, or American Society of anaethesiology (ASA) I-II
3. Stage IA2-IB1-IB2-IIA1-IIA2-IIB cervical cancer according to FIGO (International Federation of Gynecology and Obstetrics) staging.
4. Stage II, III endometrial cancer

Exclusion Criteria:

1. Non Invasive Cancer
2. Pregnancy
3. Bladder dysfunction detected prior to surgery.
4. Previous pelvic lymphadenectomy.
5. Tumour recurrence
6. Incomplete surgery, unresectable lesion.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2014-11 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Functional outcome of laparoscopic nerve sparing radical hysterectomy type III/C1 | 1 month
  Duration of postoperative catheterization untill PVR urine volume is less than 100 ml

SECONDARY OUTCOMES:
Intraoperative complications | During Surgery
  intraoperative complications
Blood loss | Day of surgery
  Amount of blood intraoperative blood loss in ml. units
Operative time | Day of surgery
  Minutes for the surgical intervention
Early postoperative complication | 30 days
  Occurence of early postoperative complication within 30 days of operation
Late postoperative complication | more than 30 days postoperative
  complications related to surgery more than 30 days postoperative
Bladder training exercise | 1 month
  Removal of urinary catheter on the 3rd day postoperative without prior bladder training exercise and measurement of PVR urine volume

CONTACTS AND LOCATIONS:
Overall Officials: Khaled Gaballa, MS.c., Principal Investigator — Assistant Lecturer of surgical oncology, Mansoura universitry; Adel Taha Denewar, M.D., Ph.D, Study Chair — Head of surgical oncology department, Mansoura oncology centre, Mansoura university; Giovanni Scambia, M.D.,Ph.D, Study Director — Head of the Department for Woman and Unborn Life Health Care- Catholic University of the Sacred Heart- Rome, Italy; Valerio Gallotta, M.D., Study Director — Department of Gynecologic Oncology,Catholic University of the Sacred Heart,Rome,Italy
Locations (2):
- Al Mansurah, Dakahlia Governorate, Egypt
- Largo Agostino Gemelli, Roma, RM, Italy